CLINICAL TRIAL: NCT03367455
Title: Interaction of Potassium Measures With Potassium Channel Genetic Variants on Diabetes Risk: The Atherosclerosis Risk in Communities (ARIC) Study and Jackson Heart Study (JHS)
Brief Title: Interaction of Potassium and Genetic Risk Variants on Diabetes Risk
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Johns Hopkins University (Other); University of Colorado, Denver (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00065581
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Diabetes
Keywords: Potassium; Genetic Variants
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARIC and JHS participants: A combined cohort of Atherosclerosis Risk in Communities (ARIC) Study and Jackson Heart Study (JHS) participants

SUMMARY:
The investigators propose to study the association of the KCNJ11 (Potassium Voltage-Gated Channel Subfamily J Member 11) polymorphisms on diabetes risk in the Atherosclerosis Risk in Communities (ARIC) and Jackson Heart Study (JHS) cohorts. The investigators also propose to test for an interaction between serum K and these genetic variants. By testing for such an interaction, it will be determined if, among participants with these genetic variants, a low-normal serum K was a stronger predictor of diabetes risk compared to those participants without these genetic variants.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Atherosclerosis Risk in Communities (ARIC) Study or Jackson Heart Study (JHS) cohorts

Exclusion Criteria:

* Had not fasted 8 or more hours for the baseline visit
* Prevalent diabetes at baseline exam
* Missing information on serum potassium
* Missing single nucleotide polymorphism (SNP) data
* Evidence of kidney dysfunction
* Race other than black/African American or white/Caucasian
* Missing other covariates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The ARIC study is a prospective cohort of 15,792 adults between the ages of 45 and 64 years at the baseline visit. Participants were recruited from four communities in the US-Forsyth County, North Carolina, Jackson, Mississippi, Minneapolis, Minnesota, and Washington County, Maryland. All participants attended an initial baseline visit between 1987-1989. JHS is a community-based, prospective cohort study of 5301 African-American adults, aged 21-95 years at the baseline visit, from the Jackson, Mississippi metropolitan area. Participants had baseline data collected between 2000 and 2004.
Sampling Method: Non-Probability Sample
Enrollment: 11812 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Associations of serum potassium and KCNJ11 variants with incident diabetes as represented by odds ratio | through study completion, mean of 8 years of follow-up
  Calculation of odds ratio will be used to represent the risk of incident diabetes associated with serum K, rs5215, and rs5219 within the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Ranee Chatterjee, MD, MPH, Principal Investigator — Duke Health

IPD SHARING:
Plan to Share IPD: No